CLINICAL TRIAL: NCT06422754
Title: THE EFFECT OF VIRTUAL REALITY APPLICATIONS ON SITTING BALANCE IN HEMIPLEGIA: A RANDOMIZED CONTROLLED STUDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-FTR-EK-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Hemiplegia
Keywords: virtual reality; hemiplegia; sitting balance
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Group (Active Comparator): The first group will receive 30 sessions of conventional exercises for 1 hour every day. In addition, the patient will be given a home program.
  Interventions: Device: Becure GmbH
- Virtual Reality Group (Active Comparator): In the second group, conventional exercises will be applied for 1 hour and 30 sessions every day. In addition to conventional exercise, this group will be enrolled in the balance game group using the Becure Balance System application and Wİ balance board for 45 minutes 5 sessions a week.
  Interventions: Device: Becure GmbH

INTERVENTIONS:
Device: Becure GmbH — Becure Balance System

SUMMARY:
Objective: The aim of this study was to investigate the effects of virtual reality application on quality of life and functionality, especially sitting balance, in hemiplegic patients.

DETAILED DESCRIPTION:
This study was planned as a single-blind randomized controlled prospective study. Patients over 18 years of age with a diagnosis of hemiplegia who applied to Gaziosmanpaşa Training and Research Hospital PTR outpatient clinic and were hospitalized in the rehabilitation service and started a rehabilitation program; will be evaluated with Modified Ashworth, Tardiue Scale, Brunstrom assessment, Stroke Specific Quality of Life Scale, Beck Anxiety Scale, Functional Independence Scale, Mini Mental State Test (MMDT), Mini Mental Test for the Uneducated, Postural Assessment Scale in Stroke Patients, Rivermead Motor Assessment Scale, Sitting Function Test, Berg Balance Scale, System Usability Scale before and after the program.

Patients who apply to the rehabilitation program will be randomly selected by closed envelope method. The first group will receive conventional rehabilitation program and home program. Conventional exercises* of the first group will be performed for 30 sessions of 1 hour every day, in addition to this, the patient will be given a home program.

In the second group, conventional exercises will be performed for 30 sessions of 1 hour every day. In addition to conventional exercises, this group will be enrolled in a balance game group using the Becure Balance System application and the WI balance board for 45 minutes 5 sessions a week.The necessary software and equipment for the virtual reality program were donated by Becure GmbH.

Both groups will be reassessed after 30 sessions. The physician performing the evaluation will be completed blindly by physiotherapists who apply the conventional exercises and the virtual reality program.

The study is a single-center clinical study using prospective data. Between 01.05.2024-01.08.2024, 36 patients are planned to be enrolled in the study.

*:Conventional exercise therapy includes range of motion, stretching, strengthening and balance exercises in patients with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Stable medical condition 2. Over 18 years of age 3. A score of 23 or above on the mini mental state test (MMDT) or the mini mental state test for the untrained (MMDT-E) 4. Within the period of 1-18 months after stroke 5. A score of 3 or 4 on the 3rd item of the Berg Balance Scale (BBS), which evaluates the balance of sitting without support (3= can sit for 2 minutes under supervision, 4= can sit safely for 2 minutes).

Exclusion Criteria:

* 1. Previous history of stroke 2. Aphasic patients in whom information exchange is not possible 3. Patients with impaired vision, hearing and vestibular system 4. Musculoskeletal and nervous system disorders other than stroke that may cause physical disability 5. Patients with a history of epilepsy 6. Cerebrovascular attack involving more than one hemisphere 7. Presence of cerebellar lesions or impaired cerebellar tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
modified ashworth scale | 1 month
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone.
Brunnstrom Stages | 1 month
  The Brunnstrom recovery stages (BRS) is a short and easily administered measure for assessing motor function.
stroke-specific quality of life | 1 month
  The QOLS was originally a 15-item instrument that measured five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation.
beck anxiety inventory | 1 month
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
The Functional Independence Measure | 1 month
  The instrument includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.
mini mental state examination | 1 month
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Postural Assessment Scale for Stroke | 1 month
  It contains 12 four-level items of varying difficulty for assessing ability to maintain or change a given lying, sitting or standing posture.
Rivermead Motor Assessment Scale | 1 month
  The Motor Assessment Scale (MAS) is a clinical assessment tool that evaluates eight areas of motor function in recovering stroke patients
function in sitting test | 1 month
  The FIST tests balance in seated position. The patient should perform items with their best posture and balance, and while moving in a seated position. The therapist will give them occasional light pushes to test for balance reactions. The therapist will make sure they won't lose their balance.
berg balance scale | 1 month
  The Berg Balance Scale is a testing tool with high validity and reliability used to measure balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Erva Kahraman, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Fergusson D, Levac D, Finestone H. Does the addition of virtual reality training to a standard program of inpatient rehabilitation improve sitting balance ability and function after stroke? Protocol for a single-blind randomized controlled trial. BMC Neurol. 2016 Mar 31;16:42. doi: 10.1186/s12883-016-0563-x. PMID 27036515
- [Background] Karasu AU, Batur EB, Karatas GK. Effectiveness of Wii-based rehabilitation in stroke: A randomized controlled study. J Rehabil Med. 2018 May 8;50(5):406-412. doi: 10.2340/16501977-2331. PMID 29620137
- [Background] Marques-Sule E, Arnal-Gomez A, Buitrago-Jimenez G, Suso-Marti L, Cuenca-Martinez F, Espi-Lopez GV. Effectiveness of Nintendo Wii and Physical Therapy in Functionality, Balance, and Daily Activities in Chronic Stroke Patients. J Am Med Dir Assoc. 2021 May;22(5):1073-1080. doi: 10.1016/j.jamda.2021.01.076. Epub 2021 Feb 24. PMID 33639116